CLINICAL TRIAL: NCT07328295
Title: Additional Effects of Thoracic Spine Mobilization Combined With Glenohumeral Joint Mobilization on Pain, Range of Motion, and Functional Disability in Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/22
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Adhesive Capsulitis
Keywords: adhesive capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic spine mobilization with Glenohumeral joint mobilization (Experimental): Participant receive Thoracic spine mobilization with Glenohumeral joint mobilization to enhance shoulder mechanics and outcomes
  Interventions: Procedure: Thoracic spine mobilization with Glenohumeral joint mobilization
- Glenohumeral joint mobilization (Active Comparator): Participant receive Glenohumeral joint mobilization only to enhance shoulder mechanics and outcomes
  Interventions: Procedure: Glenohumeral joint mobilization only

INTERVENTIONS:
Procedure: Thoracic spine mobilization with Glenohumeral joint mobilization — Thoracic spine mobilization: Central posterior-anterior (PA) oscillatory mobilizations in prone position; 30 repetitions per set, with a 1-minute rest between 2 sets.
  Glenohumeral joint mobilization: Oscillatory techniques, 2-3 oscillations per second for 30 seconds, repeated for 5 sets.
  Arms: Thoracic spine mobilization with Glenohumeral joint mobilization
Procedure: Glenohumeral joint mobilization only — Glenohumeral joint mobilization only Technique: Oscillatory mobilizations, 2-3 oscillations per second for 30 seconds, repeated for 5 sets.
  Arms: Glenohumeral joint mobilization

SUMMARY:
Adhesive capsulitis is a debilitating shoulder condition characterized by pain, restricted range of motion (ROM), and significant functional limitations. Conventional treatment primarily targets the glenohumeral joint, often neglecting the role of regional interdependence, particularly the thoracic spine's influence on shoulder mobility. Emerging evidence suggests that thoracic spine mobility plays a crucial role in optimizing shoulder mechanics, yet its therapeutic application in adhesive capsulitis remains underexplored. This study aims to investigate the additional effects of thoracic spine mobilization combined with glenohumeral joint mobilization, providing a more comprehensive rehabilitation approach to enhance pain relief, ROM, and functional outcomes.

A randomized controlled trial (RCT) will be conducted over one year at the Rehabilitation Department of Fauji Foundation Hospital (FFH) after obtaining ethical approval. Participants diagnosed with adhesive capsulitis will be selected through non-probability purposive sampling based on predefined inclusion and exclusion criteria. Subjects will be randomly assigned to either the experimental group receiving thoracic spine mobilization alongside glenohumeral joint mobilization or the control group receiving glenohumeral joint mobilization alone. Randomization will be conducted using the coin toss method and block randomization to ensure balanced subject distribution.

Outcome measures include the Numeric Pain Rating Scale (NPRS) for pain assessment, the Shoulder Pain and Disability Index (SPADI) for functional disability evaluation, and a goniometer for ROM measurement. Baseline and post-treatment scores will be statistically analyzed using SPSS to determine intervention effectiveness. By integrating thoracic spine mobilization into standard treatment, this study seeks to refine clinical rehabilitation protocols, improve functional recovery, and enhance patient outcomes. Findings may contribute to evidence-based practice, supporting the inclusion of thoracic spine mobilization in treatment guidelines for adhesive capsulitis.

DETAILED DESCRIPTION:
Adhesive capsulitis, widely known as frozen shoulder, is a progressive musculoskeletal condition characterized by shoulder pain, restricted range of motion (ROM), and marked functional limitations. Traditional treatment approaches have largely focused on mobilization techniques directed at the glenohumeral joint, aiming to reduce capsular tightness and restore movement. While this is effective to some degree, it does not fully address the concept of regional interdependence, where dysfunction in adjacent regions, particularly the thoracic spine, may influence shoulder function. The thoracic spine plays a vital role in maintaining optimal shoulder kinematics by supporting scapular positioning, facilitating overhead motion, and reducing compensatory stress on the glenohumeral joint. Stiffness or hypomobility in this region may therefore perpetuate pain and mechanical restriction in adhesive capsulitis. Treatment strategies that combine glenohumeral joint mobilization with thoracic spine mobilization have the potential to provide superior outcomes compared to conventional therapy alone. Thoracic mobilization techniques, including central and unilateral posterior-anterior glides, enhance spinal extension and rotation, indirectly improving scapular mobility and shoulder elevation. When paired with targeted glenohumeral mobilizations such as anterior, posterior, and inferior glides, patients may experience greater improvements in pain relief, ROM, and functional ability. These three variables-pain, ROM, and functional disability-are critical in determining treatment effectiveness. By incorporating thoracic mobilization into standard rehabilitation, clinicians may adopt a more holistic approach that enhances recovery, promotes long-term function, and improves the quality of life for individuals with adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* • Both male and female patients with a primary complaint of unilateral or bilateral shoulder pain

  * Pain has persisted for at least 3 to 4 months
  * Decreased shoulder ROM observed, including external shoulder rotation, abduction, internal rotation, and flexion
  * Age range between 40 to 65 years
  * Diagnosed with stage 2nd or 3rd of the disease.

Exclusion Criteria:

* • Patients if they had any shoulder pain resulting from systematic disease such as Rheumatoid Arthritis (morning stiffness > 1 hour, multiple small joints pain/swelling) Infection, Tumors, and conditions like myelopathy (Hoffman's sign).

  * Recent shoulder joint fracture/ trauma.
  * Thoracic Outlet Syndrome (Roos test).
  * The presence of Cervical radiculopathy (Spurling's test)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  Pain intensity will be checked by Numeric pain rating scale NPRS, where patient will rate pain from 0 to 10, 0 being no pain and 10 means worst pain.
Functional disability | 4 weeks
  Shoulder Pain and Disability Index (SPADI) used to assess functional disability and it is 13-question survey (5 pain, 8 disability) on a 0-100 scale, where 0 is best (no pain/difficulty) and 100 is worst (severe pain/complete disability), indicating higher scores mean greater impairment; it's interpreted by looking at general ranges (0-20 mild, 21-40 moderate, etc.) and tracking changes (a 10-20 point shift suggests clinical significance) to gauge treatment effectiveness.
Shoulder Range of Motion | 4 weeks
  Goniometer used to measure shoulder joint range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Punjab Province, Pakistan